CLINICAL TRIAL: NCT04914273
Title: Exhaled Particles in Lung Pharmacokinetics
Brief Title: Use of Exhaled Particles to Assess Lung Pharmacokinetics
Acronym: EXPLORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Prof. Dr. Jens M Hohlfeld, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21-15 EXPLORE
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Lung Pharmacokinetic
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: 1. Ingestion 2. Inhalation (Experimental): Group A is treated in the following sequence: 1. oral drug 2. inhalative drug
  Interventions: Drug: Inhalation Spray; Drug: Tablet
- Sequence B: 1. Inhalation 2. Ingestion (Experimental): Group B is treated in the following sequence: 1. inhalative drug 2. oral drug
  Interventions: Drug: Inhalation Spray; Drug: Tablet

INTERVENTIONS:
Drug: Inhalation Spray — 400 mcg salbutamol administered per metered dose inhaler
Drug: Tablet — 8 mg salbutamol administered per tablet for ingestion

SUMMARY:
This research project in humans aims at increasing the general understanding of lung pharmakokinetic by sampling exhaled particles. The central hypothesis of this study is that pharmacokinetics of Salbutamol (model drug) can be monitored in exhaled particles.

DETAILED DESCRIPTION:
The aim of the present study is to increase the general understanding of lung pharmakokinetic by systematically sampling exhaled particles at pre-specified quantities to reproduce and extent existing pilot data. For comparison, samples of blood plasma and nasal filter samples (nasosorption) will be collected for pharmakokinetic analyzes. Nasosorption will be performed to explore the possibility of detecting drug concentrations in nasal filter paper samples.

Salbutamol will be administered by inhalation and orally in a cross-over study design and both application routes shall be comparised regarding the detection of pharmakokinetic data. The aim of the study is not to generate safety or efficacy data of the selected licensed drugs. The choice of drugs is based on general considerations regarding therapy of airway diseases and the physical-chemical properties of the compounds. It is not driven by the compounds per se.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Healthy male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are:

   Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).

   Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
3. Body mass index between 18 and 32 kg/m2
4. Normal lung function with FEV1 predicted ≥ 80% and FEV1/FVC ≥ 70% at screening V1 ( or performed within 12 months prior to the screening visit at Fraunhofer ITEM and no evidence of clinical relevant abnormal findings in the lung function in the previous year before screening in the anamnesis).
5. Nonsmokers with a history of less than 1 pack year having been nonsmokers for at least the last 12 months
6. Emission of acceptable quantities of exhaled particles at screening (>200ng particle mass within 15 min)

Exclusion Criteria:

1. Any clinically relevant abnormal findings, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to asthma, chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
3. Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
4. Clinically relevant history of allergy as judged by the investigator
5. Intolerance or contraindications to salbutamol
6. Infections of the lower respiratory tract within 4 weeks before visit 1, visit 2 or visit 3. These patients can be rescreened starting from visit 1.
7. Participation in another clinical trial with an IMP 30 days or five half-lives, whichever is longer, prior to enrollment
8. History of drug or alcohol abuse
9. Risk of non-compliance with study procedures
10. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
11. Significant nasal deformity, recent nasal surgery or obstructing nasal polyps

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Salbutamol concentration assessed in exhaled particles over 5 hours after inhaled versus oral administration | Before, 0 min, 20 min, 40 min, 60 min, 120 min, 180 min, 240 min, 270 min, 300 min after drug administration

SECONDARY OUTCOMES:
Salbutamol concentration assessed in blood plasma over 5 hours after inhaled versus oral administration | Before, 0 min, 15 min, 35 min, 55 min, 75 min, 135 min, 195 min, 255 min, 285 min, 315 min after drug administration
Salbutamol concentration assessed in nasal filter samples (nasosorption) over 5 hours after inhaled versus oral administration | Before, 0 min, 15 min, 35 min, 55 min, 75 min, 135 min, 195 min, 255 min, 285 min, 315 min after drug administration
Safety and tolerability of the sampling method by assessing adverse events | Day 1 to Day 18

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz K, Biller H, Windt H, Koch W, Hohlfeld JM. Characterization of exhaled particles from the healthy human lung--a systematic analysis in relation to pulmonary function variables. J Aerosol Med Pulm Drug Deliv. 2010 Dec;23(6):371-9. doi: 10.1089/jamp.2009.0809. Epub 2010 May 25. PMID 20500095
- [Background] Schwarz K, Biller H, Windt H, Koch W, Hohlfeld JM. Characterization of exhaled particles from the human lungs in airway obstruction. J Aerosol Med Pulm Drug Deliv. 2015 Feb;28(1):52-8. doi: 10.1089/jamp.2013.1104. Epub 2014 Jun 10. PMID 24914577